CLINICAL TRIAL: NCT01333657
Title: A Prospective Study on the Diagnosis, Severity and Prognosis of Soluble Triggering Receptor Expressed on Myeloid Cells-1 in Sepsis & Related Complications
Brief Title: The Application of Soluble Triggering Receptor Expressed on Myeloid Cells-1 in Sepsis & Relevant Acute Kidney Injuries
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Lixin Xie, Pneumology Department of Chinese PLA General Hospital
Other Study IDs: 301PLAGH-20090923-001; 2009BAI86B03 (Other Grant/Funding Number: Chinese National Science & Technology Pillar Program)
Record Dates: First submitted 2011-04-07; First posted 2011-04-12 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2011-03

CONDITIONS: SIRS; Sepsis
Keywords: sTREM-1; sepsis; SIRS; blood; urine; diagnosis; prognosis
MeSH Terms: conditions — Sepsis; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- SIRS: 1. temperature >38 ℃ or <36℃;
  2. pulse rate>90 beats/min;
  3. ventilatory rate>20 breaths/min or hyperventilation with partial pressure of arterial carbon dioxide (PaCO2)<32mmHg;
  4. white blood cell count>12,000μL-1 or <4000μL-1 or >10% immature cells
- Sepsis: 1. sepsis: SIRS plus infection;
  2. severe sepsis: sepsis associated with organ dysfunction, hypoperfusion, or hypotension;
  3. septic shock: sepsis with arterial hypotension, despite adequate ﬂuid resuscitation.

SUMMARY:
Triggering receptor expressed on myeloid cells-1 is a member of the immunoglobulin superfamily of receptors that is specifically expressed on the surfaces of monocytes and neutrophils.TREM-1 expression is increased in infectious diseases and is associated with the release of soluble TREM-1 (sTREM-1).There has been demonstrated that the value of plasma sTREM-1 levels as an indicator of sepsis was superior, although other studies reported that the value of sTREM-1 for diagnosing sepsis was inferior.An increasing number of studies indicate that there are increased levels of sTREM-1 in body fluid samples for the following diseases and conditions: sepsis, pneumonia, pleural effusion, septic arthritis, meningitis, peritonitis, and uterine cavity infection.

Inflammation is now believed to play a major role in the pathophysiology of AKI. It is hypothesized that the initial insult results in morphological and/or functional changes in vascular endothelial cells and/or in tubular epithelium in sepsis models. Then, leukocytes including neutrophils, macrophages, natural killer cells, and lymphocytes infiltrate into the injured kidneys and induce the generation of inflammatory mediators. Whether urine sTREM-1 could also be detected and its significance in sepsis and AKI has not been reported yet.

The present study focused on the value of serum & urine sTREM-1 for sepsis identification, severity and prognosis assessments, and potential sepsis-related AKI. We also made comparisons between sTREM-1 and WBC counts, serum CRP, serum PCT, urine output,CC SCr, and BUN among sepsis patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female aged 18 years old and over;
2. clinically suspected infection;
3. fulfilled at least two criteria of systemic inflammatory response syndrome (a) core temperature higher than 38 °C or lower than 36 °C (b)respiratory rate above 20/min, or PCO2 below 32 mmHg (c) pulse rate above 90/min, and (d) white blood cell count greater than 12,000/μl or lower than < 4,000/μl or less than 10% of bands.

Exclusion Criteria:

Those who fulfilled one below:

* neutropenia (≤ 500 neutrophils/mm3)
* HIV infection, and
* patients or their relatives refused

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between May 2010 and March 2011, inpatients were included who were in the intensive care units (ICU) of the Department of Respiratory Disease, the Emergency Department, and the Department of Surgery of the Chinese People's Liberation Army General Hospital.
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2010-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Patients Outcome | 28 days
  The survival time of patients more than 28days is defined as survival. The survival time of patients less than 28days is defined as death.

CONTACTS AND LOCATIONS:
Overall Officials: Xie Lixin, Doctor, Study Director — Pneumology Department of chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, China

REFERENCES:
- [Derived] Su LX, Feng L, Zhang J, Xiao YJ, Jia YH, Yan P, Feng D, Xie LX. Diagnostic value of urine sTREM-1 for sepsis and relevant acute kidney injuries: a prospective study. Crit Care. 2011;15(5):R250. doi: 10.1186/cc10508. Epub 2011 Oct 24. PMID 22023777